CLINICAL TRIAL: NCT06655077
Title: Incorporating PRO Data Into RA Clinical Encounters Using Health IT
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-18282; R01HS025405 (AHRQ)
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis
Keywords: electronic dashbaord; patient reported outcomes
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control phase (No Intervention): Any patient visits that occur before the time at which clinicians are granted access to the RA PRO dashboard will be part of the control phase (usual care).
- Intervention phase (Experimental): Any patient visits that occur after the time at which clinicians are granted access to the RA PRO dashboard will be part of the intervention phase. The RA PRO dashboard will automatically launch into a new "tab" when the EHR is opened for any RA patient with at least 1 CDAI documented.
  Interventions: Other: RA PRO Dashboard

INTERVENTIONS:
Other: RA PRO Dashboard — The RA PRO Dashboard was developed by UCSF rheumatology investigators in collaboration with the UCSF SOMTech Unit. Briefly, investigators used a human-centered design approach to build a new, EHR-integrated, patient-facing visualization tool that displays RA outcome data to RA patients during clinical visits. The RA PRO dashboard was tailored for deployment at the UCSF Health's rheumatology clinic using a EHR side-car application (Salesforce). The dashboard was launched into the production environment in August 2021. With the launch, investigators integrated quality improvement, user monitoring, and lean management techniques to promote use of RA outcomes and the dashboard (for clinicians granted access) during clinical visits.
  Other Names: PACT Dashboard
  Arms: Intervention phase

SUMMARY:
The goal of this pragmatic clinical trial is to learn if a new health IT tool that was rolled out at UCSF Health rheumatology clinics (the RA PRO dashboard) can help improve the lives of individuals with rheumatoid arthritis. The RA PRO dashboard displays important outcomes for individuals with rheumatoid arthritis, including disease activity, physical functioning, and pain scores in an easy-to-read, digital interface that can be displayed on the computer screen during a clinical visit. These outcomes are tracked over time, so patients and clinicians can see changes across multiple time points. Additional features of the dashboard include displaying medication use over time and recent lab test results.

The main questions the study aims to answer are: Does displaying the dashboard during a clinical visit ...

1. reduce decisional conflict when making a medication choice?
2. improve self-efficacy in symptom management?
3. change beliefs about medications?
4. improve medication adherence?
5. improve RA outcomes such as disease activity or physical functioning?

Researchers will compare these outcomes in the patients of clinicians who have access to the RA PRO dashboard to those who do not to see if these outcomes change over time.

Clinicians with access to the dashboard may choose to share it from the computer screen with patients during the clinic visit. Participants will be asked to complete surveys as part of their routine clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis
* Visits with clinicians at UCSF Health clinic
* At least 1 CDAI score documented in UCSF EHR

Exclusion Criteria:

* Unable to read, speak, or understand English
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
SURE | Collected during routine clinical visits throughout study period; on average 3 times per year, up to 2 years.
  The SURE Test (Sure of myself; Understand information; Risk-benefit ratio; Encouragement) is a 4-item scale that measures decisional conflict in patients using a binary scale (where 0 = "no"; 1 = "yes") for a simple sum of up to 4 points. A higher score indicates greater decisional clarity.
PROMIS Short Form v1.0 - Self-Efficacy for Managing Symptoms 4a (PROMIS-SE) | Collected during routine clinical visits throughout study period; on average 3 times per year, up to 2 years.
  The PROMIS Short Form v1.0 - Self-Efficacy for Managing Symptoms 4a (PROMIS-SE) is a 4-item scale that measures self-efficacy in symptom management using a 5-point Likert-type scale (where 1 = "not at all confident"; 5 = "very confident") for a raw score range of 4 to 20, translated into T-scores with a mean of 50, and a standard deviation of 10. A higher T-score indicates greater self-efficacy.
Beliefs about Medicines Questionnaire - Specific (BMQ-Specific) | Collected during routine clinical visits throughout study period; on average 3 times per year, up to 2 years.
  The Beliefs about Medicines Questionnaire - Specific (BMQ-Specific) is comprised of two 5-item subscales that assess patients' beliefs about their need for medication to maintain health (Specific-Necessity) and their concerns about its potential negative effects (Specific-Concerns) using a Likert-type scale (1 = "strongly agree"; 5 = "strongly disagree") for a simple sum of 5 to 25 points for each subscale. Responses are used to calculate the Necessity-Concerns differential (Specific-Necessity minus Specific-Concerns) to assess patients' need for medication in comparison to their concerns. Scores range from -20 to +20, where a positive score indicates that necessity beliefs outweigh concerns.
Medication adherence | Collected during routine clinical visits throughout study period; on average 3 times per year, up to 2 years.
  Medication adherence was measured using a single item ("How many times do you think you may have missed taking your pills in the last week?"). A higher result indicates lower medication adherence.

SECONDARY OUTCOMES:
CDAI score | Collected during routine clinical visits throughout study period; on average 3 times per year, up to 2 years.
  CDAI is a validated RA disease activity outcome (range 0-76) used in a treat-to-target approach to RA treatment. It is collected routinely in the clinic by clinicians and documented in the EHR. A higher score indicates more disease activity.
PROMIS-PF10a score | Collected during routine clinical visits throughout study period; on average 3 times per year, up to 2 years.
  PROMIS-PF10a score is a validated RA functional status measure. It is collected routinely in the clinic and documented in the EHR. A higher score indicates better function.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Schmajuk, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmajuk G, Nasrallah C, Berrean B, Prugh J, Wilson C, Hamblin A, Young C, Jacobsohn L, Kay J, Li J, Kersey E, Subash M, Murray S, Yazdany J. A step-by-step roadmap for the development and deployment of an electronic health record sidecar application that tracks patient outcomes: The RA PRO dashboard. Digit Health. 2024 Oct 10;10:20552076241288739. doi: 10.1177/20552076241288739. eCollection 2024 Jan-Dec. PMID 39421306